CLINICAL TRIAL: NCT04359888
Title: A Balanced Reach Training Platform to Address Balance Disorders in Older and Neurologically Disabled Veterans
Brief Title: A Balanced Assessment and Training Protocol (BATP) to Address Balance Disorders in Older and Neurologically Disabled Veterans
Acronym: BATP
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: E3096-R; I01RX003096 (NIH)
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Older Men and Women With High Fall Risk
Keywords: Balance; Expected Balance Disturbances; Engineering Methods Related to Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MMBI: Multi-Modality Balance Intervention (MMBI) Group
  Interventions: Other: Multi-Modality Balance Intervention
- BRT Group: Balanced Reach Training Group
  Interventions: Other: Balanced Reach Training (BRT)

INTERVENTIONS:
Other: Multi-Modality Balance Intervention — Three one-hour training sessions 2-3x per week for six weeks in Multi-Modality Balance Intervention (MMBI). (See Study Design)
  Other Names: MMBI
  Groups: MMBI
Other: Balanced Reach Training (BRT) — One-hour training sessions 2-3x per week for six weeks in the Balanced Reach Training Protocol (BRTP) (See Study Design).
  Other Names: BRT
  Groups: BRT Group

SUMMARY:
Falls are by far the leading cause of accidental injury and death in older adults. The Veteran population is more severely affected by falls since it is significantly older than the overall population (45% over 65 years of age vs. 13%); and Veterans would benefit substantially more from an accurate diagnosis and treatment of fall propensity. Despite its importance, much is still unknown about the manner in which balance control is compromised by age and disease. Therapeutic interventions for people who are at risk of falling have proven to be of limited utility. Engineering methods are well suited to study and evaluate balance; but have to date been applied to overly simplified scenarios that lack the complexity to probe the musculoskeletal and neurophysiological bases for balance and falls.

The long term objective of this research, which began with a VA Rehabilitation Research & Development (RR&D) Career Development Award (CDA-2), is to develop improved directives and protocols for the diagnosis and treatment of balance-related posture and movement coordination problems. This proposal significantly advances engineering methods to address existing gaps in the diagnosis and treatment of balance impairments through the development of a Balanced Assessment and Training Protocol (BATP). The BATP continuously challenges subjects to perform reaching tasks at the limits of their balance for an extended period of time, and increases these limits as subjects demonstrate improved performance. The goal of this tool is to quantitatively assess and improve at-risk individuals' ability to maintain balance when disturbed by volitional movements of the body and its parts-an important class of balance disturbances integral to many activities of daily living that can precipitate falls. The BATP focuses on performance at and just beyond the limits of balance, unlike most such tests and training protocols that do not challenge subjects in this way. The BATP's most immediate and salient metric is the limiting boundary of standing reach; and we hypothesize that expanding this boundary, as the BATP is designed to do, will improve balance and make individuals more resistant to falls (in the context of expected balance disturbances).

Confirmation of this hypothesis could provide a new perspective on existing training protocols' modest success rates, and direction for the design of new protocols with the potential to significantly improve these rates. [Though the BATP is a training platform, we also believe that the performance metrics and analytical results produced by it can form the basis for new diagnostic measures that more reliably and precisely quantify and explain balance performance problems; and track changes in them over time.] Such diagnostic and treatment protocols would be particularly beneficial to the VA Health Care System, as it would lead to improvements in: patient throughput, quality of care, and treatment costs. Though this proposal targets the aging Veteran population, the BATP is a general tool that can aid in the diagnosis and treatment of balance disorders arising from conditions other than aging. These include obesity, diabetes (which often leads to lower extremity muscle degeneration and peripheral neuropathy), sarcopenia, vestibular disorders, and neurological disorders such as stroke. Veterans whose balance has been compromised by Traumatic Brain Injury (TBI) (whether combat-related or not) may also benefit from the BATP.

DETAILED DESCRIPTION:
Overview: This study comprises three Specific Aims (SAs): SA-1) Development of the Balanced Assessment and Training Protocol (BATP). SA-2) Assessment of the BATP's training efficacy. SA-3) Assessment of the BATP's time course of motor learning.

Methods Related to Specific Aim 1: Development of the BATP SA-1.1: Develop of the BATP's Assessment Module. The investigators will develop a BATP such that each foot's position and its associated vertical ground reaction force (used to detect stepping), as measured by the investigators' extant measurement systems, are continuously streamed to a Real Time Computing Workstation and read by the experimental control program, enabling it to monitor these quantities on an ongoing basis. The investigators will next incorporate code to establish target disk position corresponding to the subject's Limit of Balance (LoB), based on stepping. The investigators will establish LoB corresponding to seven target disk motion directions, each corresponding to a particular direction of Center of Mass (CoM) Motion. Target motion will be programmed to move unpredictably within a small circular region with center r and centerline coinciding with one of the specified directional lines. The subject then tracks the target using their dominant hand index finger until the subject (wearing a harness to guard against falling) must step to avoid a loss of balance. During this task the subject will be instructed to step rather than curtail their tracking movements when they believe they are at risk of falling. LoB in each direction is the point at which the subject steps.

The Assessment Module will record the following data to characterize performance in the tracking task

1. The values of r, , and LoB corresponding to each (Figs. 7A and 1);
2. The motion (position vs. time) of the target disk;
3. The motion of each of 15 body segments (Table 1), and the tip of the tracking finger (measured by the investigators' Vicon Motion Capture System);
4. Ground reaction forces, moments, and CoP for each foot and for both feet combined (dual Bertec force plates); All data will be saved for offline post-test processing and analyses. SA-1.2: Develop the BATP's Training Module. A single training session begins by administering the Assessment Module to establish the subject's LoB and corresponding overall target excursion amplitude, and computing the unpredictable target disk trajectory based upon it. The Training Module then presents an operator-specified number of training bouts; a single one of which consists of presenting the trajectory for the subject to track for four minutes without stepping, followed by a three minute sitting rest period. Performance data is recorded throughout the tracking period. Training bout and rest period durations can be varied (with the goal that a training session deliver 60 minutes of actual training) to optimize training efficacy and accommodate individual subject needs and capabilities. Subjects will be harnessed while performing the tracking task to guard against falling. As training progresses and the subject's performance improves, the BATP will present increasingly difficult target trajectories based upon the increased LoBs and corresponding overall target excursion amplitudes as measured by the Assessment Module at the beginning of each training session.

Methods Related to Specific Aim 2: Assessment of the BATP's training efficacy SA-2.1: Conduct the BATP and MMBI training protocols. All subject testing is performed in this Specific Aim. The investigators will screen 90 older men and women with high fall risk, enrolling 80 of these, and completing training for 68, assuming an overall 25% attrition rate.

Subjects will be randomly assigned to either the BATP or MMBI training group. Each group will receive 60 minutes of training three times per week for six weeks. BATP training is as described previously (see SA-1.2). The VA Maryland team developed an MMBI protocol for older individuals with balance and mobility disability. The program is individualized to each participant's capacity based on their balance profile and endurance level. Across the six weeks, training advances from five "fundamental" exercises that are essential for instrumental activities of daily living function to 13 exercises, as participants meet metrics for exercise safety and movement quality. Standardized progressions for each exercise advance according to the level of hand contact support required, dose (duration, sets and repetitions), intensity (movement amplitude and cadence), and multi-segmental motor challenge or complexity. The exercise cadence is adjusted up to provide greater challenge to aerobic fitness and is adjusted down to facilitate greater resistive training benefit (i.e. holding a squat longer) or to accommodate the participant's fatigue level. MMBI training will be performed in a group setting.

All subjects will be assessed with the clinical balance measures (see below) and the BATP Assessment Module at the same time points before, during, and after training (see SA-2.2).

Outcome Measures: The following "clinical measures" of balance, reach, and fall risk will be used to asses training effects induced by the BATP and MMBI.

1.Multi-Directional Reach Test 2.Falls Efficacy Scale, which assesses FoF 3.Physiological Profile Assessment (PPA) 4.Tinetti Balance Test (Balance Section) 5.Mini Balance Evaluation Systems Test (Mini-BESTest) 7.Falls experienced by each subject, as well as the conditions in which they fell, during and throughout the first year following training.

These measures will be obtained on a separate day from the BATP Assessment and Training procedures so as not to unduly fatigue the test subjects. The investigators will also employ the following BATP-based measures of balance and reach.

8.RMSE 9.RMSD-Primary Outcome Measure 10.Average SoB 11.LoB RMSD will be the investigators' primary outcome measure.

SA-2.2: Assess the training efficacy of BATP training in comparison to MMBI. Prior to training subjects will undergo double baseline tests 48 hours apart using the clinical measures and the BATP-related measures. This assessment will be repeated midway through training (three weeks after training begins), immediately post training, and six-weeks after the last training session (retention). Although the investigators include a number of clinical and BATP-related performance measures in the assessment of training efficacy, RMSD will be the investigators' primary outcome measure. The primary purpose of this study is to assess the efficacy of the BATP in improving balance. It is possible that while both the BATP and MMBI improve balance the magnitude of the difference in improvement between groups may be small. As a consequence of the relatively modest number of subjects the investigators will be testing (a result of the demands of the testing and the limited funds available to support the testing) the investigators may show no between-group difference. In order to be able to demonstrate that each intervention is efficacious, the investigators will test subjects twice at baseline and compare the change during this non-intervention period separately to the change engendered by each active intervention. The investigators' balance-related clinical measures have been shown to correlate with fall risk and fear of falling (FoF). Clinically meaningful improvements in the training group's performance based on the clinical measures will indicate that the BATP improves balance function and reduces fall risk.

The investigators will also request that subjects report any falls that they experience during the training period, and the conditions under which they fell. Once subjects have completed training the investigators will contact them monthly via e-mail, social media, or using stamped return-address post cards to obtain fall information; and follow by telephone to learn of the conditions under which they fell.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old and in good health; 60 years and older
* For ages 18-40-experienced no falls in the past year. Fall is defined as a fall that occurs under conditions that an able body individual would not fall
* For ages 60 and older-High Fall Risk or At Risk for Falling as defined by one or more of the following: Self reported fall twice or more in the past year, Self reported fear of falling, Four Square Step Test time greater than 12 seconds as determined by the study team.
* Able to perform the balanced reach task without assistive devices for 90 seconds
* Able to perform a sit-to-stand with minimal assistance and walk 10 meters without human assistance
* Adequate language and neurocognitive function to give adequate informed consent & to participate in testing and training
* Vision adequate to see a 1 inch diameter black disk against a white background at 3 feet

Exclusion Criteria:

* Any health condition that the study team deems would preclude safe completion of the BATP or MMBI
* Body Mass Index (BMI) >40
* Excessive daily alcohol consumption (>3 oz. liquor; >12 oz. wine; or >36 oz. beer) or illicit drug abuse
* For ages 60 and older-Dementia based on Montreal Cognitive Assessment (MOCA) score of less than 23 for more than 9th grade education.
* Neurological disease such as stroke, limb paralysis, Parkinson's disease, or vestibular disorders sufficient to preclude safe completion of the BATP or MMBI
* Poorly controlled hypertension (>190/105) on at least two separate occasions
* Poorly controlled type 1 or 2 diabetes (HbA1c >10)
* Recent hospitalization for severe disease or surgery (<3 month)
* Congestive heart failure or valvular dysfunction symptomatic with ordinary activities (NYHA II)
* Self-reported Pregnancy.
* Symptomatic orthostatic hypotension
* Participant has/had or currently is in a personal (romantic) relationship with any member on the study team.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the VA Maryland Health Care System (VAMHCS) Neurology, Rehabilitation, and Primary Care Clinics; the 12 hospital University of Maryland Medical System (UMMS); and the University of Maryland Rehabilitation Institute. Additional subjects will be identified using the research recruitment registries maintained by the Baltimore VA Geriatric Research Education and Clinical Center (GRECC) and UM-NIA Pepper Center. IRB-approved advertisements, mailings, and newsletters will target high fall risk older adults not currently registered for health care services at our medical centers. Participants will be chosen without regard to socioeconomic status and ethnicity.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2025-08-13 (Actual); Study Completion 2025-08-13 (Actual)

PRIMARY OUTCOMES:
Root Mean Squared Deviation between Center of Mass and Center of Base of Support (RMSD) | Assess change between base line (just prior to training) and within 24 hours of the end of training (1 week)
  Measure of Balance Capability. Root Mean Squared Deviation (RMSD) records the root mean squared distance between the ground plane projection of whole-body Center of Mass and the center of the Base of Support during performance of the balanced reach task, in centimeters. It ranges from zero to the distance from the center of the Base of Support to the boundary of the Base of Support. Larger deviations indicate better performance than smaller deviations.

SECONDARY OUTCOMES:
Multi-Directional Reach Test | Assess change between base line (just prior to training) and within 24 hours of the end of training (1 week)]
  Measures ability to lean and reach. Multi-Directional Reach Test records the distance in centimeters that one can reach in the forward, backward, rightward, and leftward directions; by bending at the waist and reaching with arm extended in each associate
Falls Efficacy Scale | Assess change between base line (just prior to training) and within 24 hours of the end of training (1 week)
  Assesses fear of falling. The Falls Efficacy Scale is a self-report questionnaire providing information on level of concern about falls for a range of activities of daily living. The questionnaire contains 16 items scored on a 1-10 point scale (1 = very confident to 10 = not very confident). The overall score is the sum of the 16 scores that are provided. Overall scores above 70 indicates a fear of falling; Lower scores are better than higher scores.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E. Barton, MD PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT04359888/ICF_000.pdf